CLINICAL TRIAL: NCT02486744
Title: Safety and Efficacy of Acthar Gel in an Outpatient Dialysis Population
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Recruitment challenges and unforseen costs to continue
Sponsor: Youngstown State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 014-2015
Record Dates: First submitted 2015-06-08; First posted 2015-07-01 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: End Stage Renal Disease
Keywords: Acthar; Dialysis; Kidney; Non-Diabetic
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 80 Units of Acthar (Active Comparator): Subjects assigned by random assignment to receive 80 Units of Acthar Gel 2x weekly for 6 months
  Interventions: Drug: Acthar Gel
- 40 Units of Acthar (Active Comparator): Subjects assigned by random assignment to receive 40 Units of Acthar Gel 2x weekly for 6 months
  Interventions: Drug: Acthar Gel

INTERVENTIONS:
Drug: Acthar Gel — Subjects will be given an injection subcutaneously 2x week for 6 months. Dosing will be randomly assigned as either 80 U or 40 U
  Other Names: repository corticotropin injection

SUMMARY:
This will be a prospective observational study of Acthar Gel in Non-Diabetic Hemodialysis [NDHD] patients receiving dialysis for ≤ 2 years. The project will aimed at providing proof-of-concept data that 80 U two times [2x] week Acthar for 6 months is a safe and effective therapy for NDHD. Effectiveness of lower dose 40 U 2X week will also be determined. Therefore the study will be a repeated measures design (Time x condition) comparison of improvement in renal function, nutritional status, quality of life and physical performance resulting from Acthar therapy.

DETAILED DESCRIPTION:
Recent reports demonstrated Acthar gel is effective to induce remission of proteinuria in the Nephrotic Syndrome patients (Bomback 2011, 2012). There are limited published reports documenting the clinical response (creatinine, proteinuria, serum albumin and cholesterol) to ACTHAR therapy in a non-diabetic hemodialysis population. In addition to renal dysfunction and high risk for mortality, individuals who receive dialysis also have decreased strength, low exercise capacity, poor physical functioning, and a low quality of life (Edgell 1996, Johansen, 2001). Strength deficits are well documented in those with End Stage Renal Disease [ESRD] (Cheema 2010, Yoda 2012). There are several reports documenting an association between strength and gait deficits and other measures of physical performance in persons with ESRD (Bohannon 1994, Fitts 1997, Segura-Orti 2011). It is well known that measures of physical performance may predict risk for fall and hospitalization in older individuals (Guralnik JM, 2000).

Deficits to physical performance may be further compounded by poor nutritional status. Persons with chronic renal disease, particularly in the context of hemodialysis or chronic renal replacement therapy, are often malnourished and/or are affected by abnormal micronutrient status (McMahon 2012). Furthermore, previous studies have shown that more than a third of acute-care, nephrology-related admissions are characterized by malnutrition (Lim 2012), and that it affects from 23% - 76% of all patients receiving hemodialysis (including outpatients)(Blumenkrantz 1980, Ikizler 1996, Pecoits-Filho 2002).

Decreased functional status and concomitant malnutrition contribute to increased hospital readmissions, prolonged length of stay (and inevitably, increased medical costs), and increased morbidity and mortality patients (Isabel 2003, Lim 2012). Given the high prevalence of these characteristics in persons with renal disease, it is important to prioritize identification of novel and effective means by which to sustain and improve the functional capability of these patients, and to maintain their nutritional status and attenuate malnutrition.

To date, there are no reports of the impact of Acthar gel therapy on renal function, strength, physical performance, nutritional status and quality of life in NDHD patients. This study will determine if Acthar gel therapy will maintain or improve overall kidney function as measured with 24 hour urine study at baseline and at the end of study period. In addition this study will determine if Acthar gel therapy will improve nutritional, physical and biochemical status in an outpatient non-diabetic hemodialysis population.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will be individuals requiring dialysis for treatment of ESRD who have had poor response to immunosuppressive strategies.
* Non-Diabetic
* Adults age 18-80

Exclusion Criteria:

* receiving hemodialysis for > 5 years
* diabetic, less than 18 years of age
* are pregnant
* have a history of cancer in the last 5 years
* have an active infection
* have recently had a myocardial infarction (within 6 weeks)
* have malignant arrhythmias, unstable angina, uncontrolled hypertension (SBP> 180 and/or DBP > 105)
* recent hospitalization (< 30 days),
* ocular disease,
* accelerated osteoporosis,
* gastrointestinal diseases (ulcerative colitis, diverticulitis, myasthenia gravis)
* any disorder that may be exacerbated by short periods of activity.
* cognitive dysfunction
* neurological deficits leading to limited ambulation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Renal Function | 6 months
  Maintain or improve renal function [Creatinine clearance and Proteinuria] by ≥ 20% , as measured by eGFR or 24 hour urine study.

SECONDARY OUTCOMES:
Hyperparathyroidism | 6 months
  Change in serum parathyroid hormone levels
Anemia | 6 months
  Change in hemoglobin levels
Inflammatory blood markers | 6 months
  Change in serum C-Reactive Protein and Creatine Kinase
Vitamin D uptake | 6 months
  Change in Vitamin D dosing requirements
Hypercalcemia | 6 months
  Change in serum calcium levels
Phosphate | 6 months
  Change in serum phosphate levels
Total Iron Binding Capacity | 6 months
  Change in Total Iron Binding Capacity in serum
Epogen Dose | 6 months
  Change in epogen dosing requirements
Fall risk | 6 months
  Timed Up and Go Test will improve
Walking endurance | 6 months
  2 minute walk distance
Gait speed | 6 months
  10 meter gait speed test
Mobility disablement risk | 6 months
  Short Performance Physical Battery
Habitual Physical Activity | 6 months
  Physical Activity Scale for the Elderly
Calf Strength | 6 months
  Heel Rise Test
Quality of life | 6 months
  Medical Outcome Study Short Form 36
Fear of Falling | 6 months
  ABC Scale [Activities-specific Balance Confidence Scale-Powell]. Scores to be above 67.
Self- Report Physical Activity | 6 months
  RAPA [Rapid Assessment of Physical Activity-Univ of Washington]
Nutritional Status | 6 months
  Body Mass Index
Lean body mass | 6 months
  Body Composition examination using Noori (2012) regression equation for lean body mass.
Caloric intake | 6 months
  Food Frequency Questionnaire (indicator of habitual intake)
Strength | 6 months
  Muscle force measures in 8 muscle groups
Nutritional Indices | 6 months
  Pre-Albumin

CONTACTS AND LOCATIONS:
Overall Officials: Erdal Sarac, MD, Principal Investigator — Renal Group
Locations (1):
- Center for Dialysis Care 3695 Stutz Drive, Canfield, Ohio, United States

IPD SHARING:
Plan to Share IPD: No